CLINICAL TRIAL: NCT04227249
Title: Three-year Recurrence Free Survival in Patients With Ultra-low-risk Endometrial Cancer Who do Not Undergo Lymph Node dissEction
Brief Title: 3 Year Recurrence Free Survival in Ultra-low-risk Endometrial Cancer
Acronym: TREE PRO
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KGOG 3021
Record Dates: First submitted 2020-01-02; First posted 2020-01-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: women who do not undergo lymph node dissection
  Interventions: Procedure: no lymph node dissection

INTERVENTIONS:
Procedure: no lymph node dissection — do not undergo lymph node dissection

SUMMARY:
To verify the safety of omission of lymph node dissection in ultra-low-risk endometrial cancer (KGOG criteria), we examine the survival of women with ultra-low-risk endometrial cancer who do not undergo lymph node dissection

ELIGIBILITY:
Inclusion Criteria:

* endometrioid type
* anticipated surgery omitting lymph node dissection for endometrial cancer
* pelvis MRI, CA125 - satisfying KGOG criteria
* no distant metastasis
* age 19 or more

Exclusion Criteria:

* other cancer within 5 yr
* previous hysterectomy
* previous therapy for endometrial cancer

Min Age: 19 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: endometrial cancer with ultra-low risk for lymph node metastasis
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
3 year recurrence free survival | 3 year since surgery
  3 year recurrence free survival

SECONDARY OUTCOMES:
5 year recurrence free survival | 5 year since surgery
  5 year recurrence free survival
5 year overall survival | 5 year since surgery
  5 year overall survival
surgery time | surgery visit
  from surgery start to end
change of Functional Assessment of Cancer Therapy - General (FACT G) score from baseline | baseline - 1week - 5week - 3month - 6month
  functional assessment of cancer therapy - general
change of Gynecologic Cancer Lymphedema Questionnaire - Korean (GCLQ-K) score from baseline | baseline - 5week - 6month - 12month - 18month - 24month - 36month - 48month - 60month
  gynecologic cancer lymphedema questionnaire - Korean
change of Female Sexual Function Index (FSFI) score from baseline | baseline - 6month - 12month - 24month - 36month - 48month - 60month
  female sexual function index
length of stay | surgery visit
  from admission to discharge
transfusion | surgery visit
  amount of transfusion
hemoglobin decline | surgery visit
  change of hemoglobin level from baseline to postoperative lowest level
surgery complication | surgery visit
  any surgery complications observed

IPD SHARING:
Plan to Share IPD: No